CLINICAL TRIAL: NCT03126227
Title: Real-World AR101 Market-Supporting Experience Study in Peanut-Allergic Children Ages 4 to 17 Years (RAMSES)
Brief Title: Real-World AR101 Market-Supporting Experience Study in Peanut-Allergic Children (RAMSES)
Acronym: RAMSES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARC007
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen; CPNA (Characterized Peanut Allergen); OIT (oral immunotherapy); Peanut Allergy; Peanut-Allergic Children; Desensitization; ARC007; Characterized Oral Desensitization Immunotherapy (CODIT™)
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: 2:1 randomization to AR101 or placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR101 Powder Provided in Capsules (Active Comparator): Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
  Interventions: Biological: AR101
- Placebo powder (Placebo Comparator): Placebo formulation in pull-apart capsules containing only excipients color-matched to AR101 study product.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AR101 — AR101 powder provided in capsules
  Arms: AR101 Powder Provided in Capsules
Biological: Placebo — Placebo powder provided in capsules
  Arms: Placebo powder

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled safety study of AR101 using the characterized oral desensitization immunotherapy (CODIT™) regimen in peanut-allergic children.

DETAILED DESCRIPTION:
The primary objective is to assess the safety and tolerability of AR101 when used in a CODIT™ regimen for approximately 6 months in peanut-allergic children children aged 4 to 17 years, inclusive.

ELIGIBILITY:
Key Inclusion Criteria:

* Ages 4 to 17 years, inclusive
* History of physician-diagnosed peanut allergy that includes allergic signs and symptoms within two hours of known oral exposure to peanut
* Mean peanut wheal diameter on SPT of at least 8mm and elevated psIgE of at least 14 kUA/L at screening
* Written informed consent from the subject's parent/guardian
* Written assent from the subject as appropriate (per local regulatory requirements)
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* Subjects in whom the clinical diagnosis of peanut allergy is uncertain
* Severe or uncontrolled asthma
* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* History of severe or life-threatening episode of anaphylaxis or anaphylactic shock within 60 days of screening
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia or recurrent gastrointestinal symptoms of undiagnosed etiology
* History of a mast cell disorder, including mastocytosis, urticaria pigmentosa, chronic idiopathic or chronic physical urticaria beyond simple dermatographism (e.g., cold urticaria, cholinergic urticaria), and hereditary or idiopathic angioedema
* Any other condition that, in the opinion of the Investigator, precludes participation for reasons of safety

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 506 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Chair — Aimmune Therapeutics, Inc.
Locations (67):
- United States (62):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Jonathan Corren, M.D., Inc., Los Angeles, California
  - Children's Hospital Los Angeles, Division of Clinical Immunology and Allergy, Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Sean N. Parker Center for Allergy Research, LPCH at El Camino Hospital, Mountain View, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, A.P.C, San Diego, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Asthma & Allergy Associates, PC, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Colorado Allergy & Asthma Centers, Denver, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Sher Allergy Specialists - Center for Cough, Largo, Florida
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - University of South Florida Asthma, Allergy, and Immunology Clinical Research Unit, Tampa, Florida
  - Atlanta Allergy & Asthma Clinic, PA, Marietta, Georgia
  - Idaho Allergy and Research, Eagle, Idaho
  - Ann & Robert H. Lurie's Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medicine, Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - University of Iowa, Iowa City, Iowa
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Johns Hopkins Hospital, Pediatric Clinical Research Unit, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System / Michigan Medicine, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - Children's Mercy on Broadway, Kansas City, Missouri
  - Nebraska Medical Research Institute, Inc., Bellevue, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Northwell Health System, Great Neck, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - National Allergy and Asthma Research, LLC, Charleston, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Columbia Asthma & Allergy Clinic, Clackamas, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, Portland, Oregon
  - Children's Hospital of Philadelphia: Allergy/Immunology, Philadelphia, Pennsylvania
  - Dell Children's Medical Group / Allergy, Asthma & Immunology Clinic, Austin, Texas
  - Children's Health, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - ASTHMA Inc. Clinical Research Center, Seattle, Washington
- Canada (5):
  - Triple A Lab (Hamilton Allergy), Hamilton, Ontario
  - McMaster University Medical Center, Hamilton, Ontario
  - Cheema Research Inc. (CRI), Mississauga, Ontario
  - Ottawa Allergy Research Corp., Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Started | 338 | 168
Completed | 260 | 158
Not Completed | 78 | 10
Not completed — Adverse Event | 43 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 19 | 3
Not completed — Discontinued due to early termination and continuation in follow-on study due to study closure | 8 | 1
Not completed — Lack of dosing compliance | 2 | 0
Not completed — Did not meet eligibility criteria subsequent to enrollment | 2 | 0
Not completed — Scheduling conflict | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 506 subjects were enrolled. However, only 505 subjects were included in the intent-to-treat (ITT) population. The ITT Population includes all subjects who received at least one dose of randomized study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder | Total
Number analyzed (Participants) | 337 | 168 | 505
Age, Continuous [Median (Full Range); unit: years] | 9.0 [4 to 17] | 9.5 [4 to 17] | 9.0 [4 to 17]
Age, Customized [Count of Participants; unit: Participants]
  4-11 years | 226 | 114 | 340
  12-17 years | 111 | 54 | 165
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 66 | 185
  Male | 218 | 102 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 8 | 27
  Not Hispanic or Latino | 318 | 159 | 477
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 39 | 25 | 64
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 11 | 4 | 15
  White | 245 | 113 | 358
  More than one race | 33 | 11 | 44
  Unknown or Not Reported | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment Emergent Adverse Events, Including Serious Adverse Events
Description: Frequency of Treatment Emergent Adverse Events, including Serious Adverse Events, during the overall study period.
  Treatment-emergent adverse events were defined as adverse events with onset after the first dose of study product.
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants
  Subjects with at least 1 AE | 334 | 159
  Mild AE | 171 | 110
  Moderate AE | 151 | 47
  Severe AE | 11 | 1
  Life Threatening AE | 1 | 0
  Death | 0 | 1
  Subjects with at least 1 serious adverse event | 2 | 2

2. Secondary Outcome: Frequency of Premature Discontinuation of Dosing Due to Adverse Events
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 41 | 5

3. Secondary Outcome: Frequency of Premature Discontinuation of Dosing Due to Chronic/Recurrent Gastrointestinal Adverse Events
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 20 | 0

4. Secondary Outcome: Proportion of Chronic/Recurrent Gastrointestinal Adverse Events Resolving <2, Between 2-4, Between 4-12, and ≥ 12 Weeks Following Discontinuation of Dosing
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment.
  Number of participants analyzed: subjects who discontinued dosing due to chronic/recurrent gastrointestinal adverse events.
  None of the subjects in Placebo group discontinued dosing due to chronic/recurrent gastrointestinal adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 20 | 0
Participants
  < 2 weeks | 17 | 0
  2-4 weeks | 2 | 0
  4-12 weeks | 0 | 0
  ≥ 12 weeks | 0 | 0
  Unknown | 1 | 0

5. Secondary Outcome: Frequency of Allergic Hypersensitivity Adverse Events Normalized for Duration of Treatment
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Number; unit: number of events
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
number of events
  Throat irritation | 1434 | 51
  Abdominal pain | 1184 | 83
  Abdominal discomfort | 911 | 65
  Nausea | 557 | 26
  Pruritus | 510 | 106
  Abdominal pain upper | 374 | 31
  Oral pruritus | 361 | 6
  Tongue pruritus | 305 | 5
  Sneezing | 296 | 41
  Vomiting | 266 | 14
  Urticaria | 251 | 117
  Cough | 195 | 64
  Lip pruritus | 170 | 0
  Rhinorrhoea | 164 | 51
  Paraesthesia oral | 159 | 39
  Rash | 139 | 62
  Nasal congestion | 127 | 47
  Throat tightness | 100 | 3
  Headache | 56 | 10
  Diarrhoea | 52 | 15
  Erythema | 51 | 20
  Anaphylactic reaction | 44 | 9
  Wheezing | 41 | 6
  Flushing | 37 | 10
  Eye pruritus | 34 | 13

6. Secondary Outcome: Frequency of Anaphylaxis as Defined in the Protocol
Description: Anaphylaxis is likely when any 1 of the 3 following sets of criteria is fulfilled:
  1. Acute onset of an illness (minutes to hours) with involvement of: (a) Skin/mucosal tissue (eg, generalized hives, itch/flush, swollen lips/tongue/uvula); AND (b) Airway compromise (eg, dyspnea, stridor, wheeze/bronchospasm, hypoxia, reduced PEFR); AND/OR (c) Reduced BP or associated symptoms (eg, hypotonia, syncope, incontinence).
  2. Two or more of the following that occur rapidly after exposure to the allergen (minutes to hours): (a) Skin/mucosal tissue; (b) Airway compromise; (c) Reduced BP or associated symptoms; (d) Persistent GI symptoms (eg, nausea, vomiting, crampy abdominal pain).
  3. Reduced BP after exposure to the allergen (minutes to hours). Infants and children: low systolic BP (age-specific) or > 30% drop in systolic BP; Adults: systolic BP < 90 mm Hg or > 30% drop from their baseline.
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 36 | 9

7. Secondary Outcome: Frequency of Epinephrine Use as Rescue Medication
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 37 | 9

8. Secondary Outcome: Frequency of Accidental Ingestion of Peanut and Other Allergenic Foods
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 26 | 31

9. Secondary Outcome: Change of Asthma Control Using the Asthma Control Test (ACT) Questionnaire Total Score From Baseline to Interim (80 mg), End of Up-Dosing (300 mg) and Study Exit, Ages 4-11
Description: The Asthma Control Test (ACT) Questionnaire ACT for subjects aged 4-11 years included 4 questions for the subject and 3 questions for the parent; the total score (sum of 7 questions) ranged from 0 (worst control) to 27 (total control)
Time Frame: Baseline, Interim dose (approx. 10 weeks), End of Up-Dosing (20 to 40 weeks), Study Exit (14 days after End of Up-Dosing, usually approx. 6 months)
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment (included subjects ages 4-11 only).
  The ACT questionnaire was not completed by all subjects and/or parents at all protocol-defined points of collection.
Measure: Mean (Standard Deviation); unit: Change in ACT total score from baseline
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 226 | 114
Change in ACT total score from baseline
  Baseline: number analyzed (Participants) | 100 | 46
  Baseline | 23.9 (2.57) | 23.7 (2.93)
  Interim (80 mg) visit: number analyzed (Participants) | 67 | 42
  Interim (80 mg) visit | 24.2 (2.52) | 23.7 (3.47)
  End of Up-Dosing (300 mg) Visit: number analyzed (Participants) | 64 | 39
  End of Up-Dosing (300 mg) Visit | 24.2 (2.63) | 23.8 (3.55)
  Study Exit: number analyzed (Participants) | 63 | 38
  Study Exit | 24.0 (3.03) | 24.5 (3.50)
  Change from Baseline to Interim (80 mg) Visit: number analyzed (Participants) | 67 | 42
  Change from Baseline to Interim (80 mg) Visit | 0.3 (2.54) | 0.2 (2.93)
  Change from Baseline to End of Up-Dosing (300 mg) Visit: number analyzed (Participants) | 64 | 39
  Change from Baseline to End of Up-Dosing (300 mg) Visit | 0.5 (3.08) | 0.4 (2.61)
  Change from Baseline to Early Discontinuation / Study Exit: number analyzed (Participants) | 63 | 38
  Change from Baseline to Early Discontinuation / Study Exit | 0.3 (3.29) | 0.7 (2.76)

10. Secondary Outcome: Change of Asthma Control Using the Asthma Control Test (ACT) Questionnaire Total Score From Baseline to Interim (80 mg), End of Up-Dosing (300 mg) and Study Exit, Ages 12-17
Description: The Asthma Control Test (ACT) Questionnaire ACT for subjects aged 12-17 years consisted of 5 questions, and the total score (sum of 5 questions) ranged from 5 (worst control) to 25 (total control).
Time Frame: as for outcome 9
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment (included subjects ages 12-17 only).
  The ACT questionnaire was not completed by all subjects and/or parents at all protocol-defined points of collection.
Measure: Mean (Standard Deviation); unit: Change in ACT total score from baseline
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 111 | 54
Change in ACT total score from baseline
  Baseline: number analyzed (Participants) | 65 | 26
  Baseline | 22.8 (2.40) | 22.9 (3.05)
  Interim (80 mg) visit: number analyzed (Participants) | 50 | 21
  Interim (80 mg) visit | 23.0 (2.69) | 23.1 (2.90)
  End of Up-Dosing (300 mg) Visit: number analyzed (Participants) | 39 | 20
  End of Up-Dosing (300 mg) Visit | 23.7 (1.73) | 23.2 (2.13)
  Study Exit: number analyzed (Participants) | 40 | 20
  Study Exit | 23.8 (1.74) | 22.6 (2.63)
  Change from Baseline to Interim (80 mg) Visit: number analyzed (Participants) | 50 | 21
  Change from Baseline to Interim (80 mg) Visit | 0.3 (2.72) | 0.2 (2.93)
  Change from Baseline to End of Up-Dosing (300 mg) Visit: number analyzed (Participants) | 39 | 20
  Change from Baseline to End of Up-Dosing (300 mg) Visit | 0.9 (1.92) | 0.5 (3.10)
  Change from Baseline to Early Discontinuation / Study Exit: number analyzed (Participants) | 40 | 20
  Change from Baseline to Early Discontinuation / Study Exit | 0.7 (1.68) | -0.2 (2.71)

11. Secondary Outcome: Frequency of Adverse Events That Led to Early Withdrawal
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of randomized study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
Number analyzed (Participants) | 337 | 168
Participants | 36 | 5

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder
All-Cause Mortality (participants affected / at risk) | 0/337 | 1/168
Serious Adverse Events (participants affected / at risk) | 2/337 | 2/168
Other Adverse Events (participants affected / at risk) | 334/337 | 159/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 Powder Provided in Capsules (N=337) | Placebo Powder (N=168)
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia mycoplasma (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 — Death due to traumatic brain injury sustained in motor vehicle accident
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 Powder Provided in Capsules (N=337) | Placebo Powder (N=168)
Abdominal pain (Gastrointestinal disorders) | 177 | 34
Abdominal discomfort (Gastrointestinal disorders) | 137 | 27
Vomiting (Gastrointestinal disorders) | 130 | 28
Nausea (Gastrointestinal disorders) | 114 | 20
Abdominal pain upper (Gastrointestinal disorders) | 75 | 24
Oral pruritus (Gastrointestinal disorders) | 50 | 5
Paraesthesia oral (Gastrointestinal disorders) | 46 | 9
Diarrhoea (Gastrointestinal disorders) | 43 | 19
Lip pruritus (Gastrointestinal disorders) | 36 | 1
Tongue pruritus (Gastrointestinal disorders) | 34 | 3
Dyspepsia (Gastrointestinal disorders) | 26 | 3
Lip swelling (Gastrointestinal disorders) | 21 | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 155 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 110 | 38
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 80 | 31
Sneezing (Respiratory, thoracic and mediastinal disorders) | 67 | 21
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 65 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 49 | 31
Wheezing (Respiratory, thoracic and mediastinal disorders) | 42 | 11
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 34 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 125 | 41
Urticaria (Skin and subcutaneous tissue disorders) | 89 | 36
Rash (Skin and subcutaneous tissue disorders) | 40 | 27
Erythema (Skin and subcutaneous tissue disorders) | 23 | 10
Upper respiratory tract infection (Infections and infestations) | 75 | 50
Nasopharyngitis (Infections and infestations) | 37 | 23
Influenza (Infections and infestations) | 29 | 9
Viral infection (Infections and infestations) | 22 | 12
Pharyngitis streptococcal (Infections and infestations) | 20 | 10
Gastroenteritis viral (Infections and infestations) | 16 | 14
Pyrexia (General disorders) | 63 | 29
Chest discomfort (General disorders) | 20 | 1
Headache (Nervous system disorders) | 91 | 44
Eye pruritus (Eye disorders) | 25 | 12
Anaphylactic reaction (Immune system disorders) | 36 | 9
Ear pruritus (Ear and labyrinth disorders) | 20 | 3
Flushing (Vascular disorders) | 26 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03126227/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03126227/SAP_001.pdf